CLINICAL TRIAL: NCT05124912
Title: REMASTer: REcurrent Brain Metastases After SRS Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Monteris Medical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REMASTer
Record Dates: First submitted 2021-10-26; First posted 2021-11-18 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Brain Metastases; Radiation Necrosis; Recurrent Tumor; Recurrent Metastases
Keywords: Laser Interstitial Thermal Therapy; Stereotactic Radiosurgry; LITT; SRS; Radiation Necrosis; Brain Metastases
MeSH Terms: conditions — Brain Neoplasms; Recurrence; Neoplasm Metastasis | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Recurrent Tumor (Other): Receives Laser Interstitial Thermal Therapy (LITT) followed by surveillance or Receives Laser Interstitial Thermal Therapy (LITT) followed by hypofractionated radiation therapy (RT).
  Interventions: Procedure: Radiation Therapy; Procedure: Laser Interstitial Thermal Therapy
- Radiation Necrosis (Other): Receives Laser Interstitial Thermal Therapy (LITT) and best medical management with steroids or Receives best medical management with steroids.
  Interventions: Drug: Steroid Therapy; Procedure: Laser Interstitial Thermal Therapy

INTERVENTIONS:
Procedure: Radiation Therapy — Post-op hypofractionated therapy or no radiation therapy
  Arms: Recurrent Tumor
Drug: Steroid Therapy — Best medical management with steroid therapy
  Arms: Radiation Necrosis
Procedure: Laser Interstitial Thermal Therapy — Minimally invasive technique to necrotize intracranial lesions using the NeuroBlate® System (NBS)

SUMMARY:
Randomized, post-market multi-center study investigating the efficacy of two sets of treatment algorithms in brain metastases (BM) patients at the time of first intervention for radiographic progression after stereotactic radiosurgery (SRS), with or without surgery.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

1. Patients with radiographically proven (by gadolinium-enhanced [Gd-] MRI) parenchymal brain metastases from histologically confirmed non-central nervous system (CNS) cancer.
2. Patients with a "targetable", bidimensionally-measurable, intracranial lesion that is radiographically recurrent after previous treatment with SRS +/- surgery (craniotomy or LITT). To classify a lesion as radiographically progressive, the lesion must demonstrate a ≥ 25% increase in size following treatment based on the Neuro-Oncology Criteria of Tumor Response for CNS Tumors. To be "targetable" for this study, the lesion should be coverable through a planned single LITT trajectory and thus have a maximum perpendicular diameter (perpendicular to the laser trajectory) of 3 cm. An intra-operative decision to utilize two trajectories is acceptable and patient may remain on study.
3. Patient must be at least 3 months post initial SRS treatment of the target lesion
4. Target lesion must be amenable to undergo surgical biopsy and LITT treatment as determined by the treating neurosurgeon.
5. Frozen pathology diagnosis must be attainable.
6. Patient must be symptomatically stable for a minimum of 3 days prior to the procedure date on a on a max total daily steroid dose equivalent to 4mg of Dexamethasone.
7. ≥18 years of age
8. KPS ≥70
9. Patient is able and willing to complete study requirements
10. Patients with adequate hematologic parameters (all tests to be performed within <4 weeks of biopsy):

    1. ANC ≥ 1.5 X 109/L
    2. Platelet count ≥ 100 x 109/L
11. Blood chemistry laboratory value for serum creatinine < 1.5 x ULN (test to be performed within <4 weeks of biopsy)
12. Female patients must have a negative serum pregnancy test at screening. (Not applicable to patients with bilateral oophorectomy and/or hysterectomy or to those patients who are postmenopausal)
13. All patients of reproductive potential must agree to use an effective method of contraception during the study
14. Patients must be accessible for follow-up

Exclusion Criteria:

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Patients with greater than 3 progressing lesions at time of enrollment. To classify as a radiographically progressive, lesion must demonstrate a ≥ 25% increase in size following treatment based on the RANO criteria. Of note, there is no exclusion for total number of metastases. However, only one lesion can be selected to be the targeted lesion and this lesion alone may be ablated during the study procedure.
2. Patients with concomitant newly diagnosed intracranial metastases (concurrent with the targetable radiographically progressive lesion), as these will require prioritized and different treatment approaches.
3. Prior bevacizumab use within 4 weeks of study initiation
4. Patients with additional concurrent malignancies requiring active treatment, except non-melanoma skin cancer, or in-situ cancer of the cervix
5. Patients with a serious active infection or other serious underlying medical conditions that would impair the ability of the patient to complete the protocol related QOL questionnaires and cognition assessments
6. Inability to tolerate or contraindication to steroid therapy (i.e., dexamethasone)
7. Deemed ineligible or unable to tolerate SRS therapy by treating neurosurgeon and/or radiation oncologist
8. Patients with any condition that would prohibit them from undergoing a surgical procedure, at the discretion of the treating physician team
9. Patients unwilling or unable to give consent for participation
10. Patients unable to comply with study requirements
11. Patients with diffuse leptomeningeal disease
12. Patients with rapidly progressing extracranial disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 261 (Estimated)
Dates: Start 2022-05-10 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Progressive Disease Cohort | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
  Determine the effectiveness of LITT using the NeuroBlate® System with or without repeat SRS on recurrent brain metastases, as measured by freedom from local progression.
Radiation Necrosis Cohort | Assessed for a three month period from time of randomization to steroid freedom without escalation of care.
  Determine the effectiveness of LITT using the NeuroBlate System versus standard medical management as measured by time to steroid independence without escalation of care, measured in days from LITT procedure, defined as freedom from steroids for a period of four weeks without escalation of care.

SECONDARY OUTCOMES:
Progressive Disease Cohort: Overall Survival | Compare treatment approaches with respect to overall survival, defined as time from study biopsy to death or study exit, up to 24 months.
  Compare treatment approaches with respect to overall survival.
Radiation Necrosis Cohort: Freedom from Local Progression (FFLP) or Neurological Death | Compare treatment approaches with respect to overall survival, defined as time from study biopsy to death or study exit, up to 24 months
  Compare treatment approaches with respect to FFLP or neurologic death

CONTACTS AND LOCATIONS:
Overall Officials: Peter Fecci, MD, Principal Investigator — University of Colorado, Denver
Locations (9):
- United States (9):
  - UCLA, Los Angeles, California
  - University of Chicago, Chicago, Illinois
  - University of Maryland, Baltimore, Maryland
  - WashU, St Louis, Missouri
  - Duke University Hospital, Durham, North Carolina
  - Wake Forest Baptist Medical Center, Winston-Salem, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Kettering Health, Kettering, Ohio
  - Medical College of Wisconsin, Milwaukee, Wisconsin